CLINICAL TRIAL: NCT03600714
Title: Treatment of Chronic Delta Hepatitis With Lonafarnib, Ritonavir and Lambda Interferon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180123; 18-DK-0123 (Other: NIH Clinical Center)
Record Dates: First submitted 2018-07-25; First posted 2018-07-26 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Liver Disease; Hepatitis D
Keywords: Hepatitis D; Hepatitis D Virus; Cirrhosis
MeSH Terms: conditions — Liver Diseases; Hepatitis D; Fibrosis | interventions — lonafarnib; Ritonavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Treatment with Lonafarnib, Ritonavir, and Peginterferon lambda
  Interventions: Drug: Peg-interferon lambda; Drug: Lonafarnib; Drug: Ritonavir

INTERVENTIONS:
Drug: Peg-interferon lambda — Peg-interferon Lambda is a covalent conjugate of human recombinant non- pegylated interferon (IFN) lambda and a 20-kDa linear pegylated (PEG) chain.
Drug: Lonafarnib — Oral prenylation inhibitor
Drug: Ritonavir — Booster of lonafarnib action

SUMMARY:
Background:

Infection with hepatitis D virus leads to a chronic liver disease with no effective treatment. Lonafarnib has improved hepatitis D virus levels in blood, but the medication still needs more research. Ritonavir makes other drugs more effective and is used with lonafarnib to make it more effective. Lambda interferon stimulates the body s response to viruses. Researchers want to see if combining these drugs fights hepatitis D and helps the liver.

Objectives:

To see if combining lonafarnib, ritonavir, and lambda interferon is safe and effective to treat chronic hepatitis D infection.

Eligibility:

Adults at least 18 years old with chronic hepatitis D infection

Design:

Participants will be screened with a physical exam, medical history, and blood and urine tests.

Throughout the study, all participants will:

* Follow rules for medicine, food, and contraception
* Take hepatitis B medicine
* Have weight checked
* Have routine blood and urine tests
* Give stool samples
* Female participants will have pregnancy tests.

Participants will have 3 visits before treatment. They will repeat screening tests and have a heart test and liver scan.

Participants will have a 5-day inpatient stay. They will:

* Baseline blood and urine tests
* Have eye tests
* Answer health questions
* Have a liver sample taken and liver blood pressure measured. Participants will be sedated.
* Have reproductive tests
* Start the study drugs and have blood draws

Over 24 weeks of treatment, participants will:

-Take 2 study drugs by mouth every day and 1 as a weekly injection

DETAILED DESCRIPTION:
Chronic delta hepatitis is a serious form of chronic liver disease caused by infection with the hepatitis D virus (HDV), a small RNA virus that requires farnesylation of its major structural protein (HDV antigen) for replication. Based on previous and ongoing clinical trials demonstrating effectiveness against HDV, we propose to treat 26 adult patients with chronic delta hepatitis using the combination of the farnesyltransferase inhibitor (FTI) lonafarnib (LNF), the protease inhibitor ritonavir (RTV) and peginterferon lambda-1a(lambda). In this phase 2a open label study, the safety and antiviral effects of triple therapy with LNF, RTV and lambda for a period of 6 months. After dosing, all patients will be monitored for 24 weeks off therapy. Nucleos(t)ide analogue therapy will be instituted/continued during this study to prevent the possibility of hepatitis B virus (HBV) reactivation/flare for the duration of participation in this clinical trial. Patients with quantifiable HDV RNA in serum will be enrolled. At each clinic visit, patients will be questioned about side effects, symptoms and quality of life, undergo focused physical examination, and have blood drawn for complete blood counts, HDV RNA, and routine liver tests (including alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, direct and total bilirubin, and albumin). At the end of the treatment, patients will be admitted to the clinical center and will undergo repeat liver biopsy and hepatic venous pressure gradient (HVPG) measurements, repeat physical examination, assessment of symptoms (using a symptom scale questionnaire), complete blood counts, routine liver tests, and hepatitis B and D viral markers. The primary therapeutic endpoint will be a decline of HDV RNA viral titer of 2 logs at the end of therapy. The primary safety endpoint will be the ability to tolerate the drugs at the prescribed dose for the full course of therapy. This clinical trial is designed as a phase 2a study assessing the antiviral activity, safety and tolerance of fixed doses of lonafarnib, ritonavir and peginterferon lambda.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 18 years or above, male or female.
* Presence of anti-HDV in serum.
* Presence of quantifiable HDV RNA in serum at three time pre-treatment points with a mean HDV RNA level >2 log10 above the lower limit of quantification (LLOQ) of the HDV RNA assay.
* Demonstration of chronicity as evidenced by the presence of HDV RNA in serum for >/= 6 months, or presence of Anti-HDV antibody >/= 6months.

EXCLUSION CRITERIA:

* Decompensated liver disease, defined by bilirubin >4mg/dL, albumin <3.0 gm/dL, prothrombin time >2 sec prolonged, or history of bleeding esophageal varices, ascites or hepatic encephalopathy. Laboratory abnormalities that are not thought to be due to liver disease may not necessarily require exclusion. Patients with ALT levels greater than 1000 U/L (>25 times ULN) will not be enrolled but may be followed until three determinations are below this level. Patients with an absolute neutrophil count <1000/dL and platelets <75,000/dL will be excluded from the study as well.
* Pregnancy, active breast-feeding, or inability to practice adequate contraception, in women of childbearing potential or in partners of such women. Adequate contraception is defined as vasectomy in male sexual partners of female participants, tubal ligation in women, or use of two contraceptive methods such as condoms and spermicide combination with an intrauterine device or Depo-Provera, or Norplant.
* Significant systemic or major illnesses other than liver disease, including, but not limited to, congestive heart failure, renal failure (eGFR <50 ml/min), organ transplantation, serious psychiatric disease or depression (only if felt to be at high risk by the NIH psychiatric consultation service), or active coronary artery disease.
* Systemic immunosuppressive therapy within the previous 2 months before enrollment.
* Evidence of another form of liver disease in addition to viral hepatitis (for example autoimmune liver disease, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson disease, alcoholic liver disease, ongoing drug induced liver disease, nonalcoholic steatohepatitis (but not steatosis), hemochromatosis, or alpha-1-antitrypsin deficiency).
* Active substance abuse, such as alcohol, inhaled or injection drugs within the previous year.
* Evidence of hepatocellular carcinoma. This will be determined on the basis of imaging with ultrasound/ CT scan or MRI performed a maximum of 6 months prior to enrollment. Elevated alpha fetoprotein (AFP) levels will be evaluated clinically and further imaging may be performed if felt necessary.
* Evidence of concurrent hepatitis C infection with positive serum hepatitis C virus (HCV) RNA.
* Any experimental therapy or pegylated interferon therapy within 6 months prior to enrollment.
* Active, serious autoimmune disease such as systemic lupus erythematosus, ulcerative colitis, Crohn s disease or rheumatoid arthritis, that is in the opinion of the investigators might be exacerbated by therapy with lambda interferon. This will be evaluated at baseline and during follow-up laboratory testing (including blood and urine studies) in addition to described symptoms at each outpatient visit.
* Diagnosis of malignancy in the five years prior to the enrollment with exception granted to superficial dermatologic malignancies.
* Evidence of HIV co-infection; HIV 1/2 antibody positivity on serum testing.
* Concurrent usage of statins as these drugs inhibits mevalonate synthesis, which reduces protein prenylation.
* Concurrent usage of moderate and strong CYTOCHROME P-450 CYP3A (CYP3A) inhibitors and inducers.
* Concurrent usage of alpha 1 adrenoreceptor antagonist, antiarrhythmic, pimozide, sildenafil, sedative and hypnotics, ergot and St. John s Wort due to possible effect of ritonavir on hepatic metabolism of these drugs resulting in potentially life-threatening side effects.
* Clinically significant baseline EKG abnormalities such as corrected QT (QTc) interval >450 ms and/or prolonged PR interval.
* Uncontrolled elevated triglycerides (>500 mg/dL). Patients on lipid lowering therapy other than statins will be eligible for this study.
* History of pancreatitis from causes other than gallstone pancreatitis. Subjects with a baseline amylase and/or lipase level >3 ULN will be excluded from the study.
* Inability to understand or sign informed consent.
* Any other condition, which in the opinion of the investigators would impede the patient s participation or compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Koh, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-DK-0123.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Patients were treated with lonafarnib 50 mg orally twice daily, ritonavir 100 mg orally twice daily and lambda 180 mcg subcutaneously weekly for 24 weeks
Period: Overall Study
Arm/Group | Treatment
Started | 26
Completed | 25
Not Completed | 1
Not completed — Out of country and could not return for post-treatment visits | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (8.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Decline of Hepatitis D Virus (HDV) RNA Viral Titer of >2 Logs
Description: Decline of HDV RNA viral titer of >2 logs from baseline at 24 weeks of therapy
Time Frame: Baseline and 24 weeks
Population: Three participants who discontinued treatment before 24 weeks did not have HDV RNA measured at 24 weeks. They were seen at post-treatment visits
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 23
Participants | 18

2. Primary Outcome: Number of Participants Who Discontinue Medication
Description: Discontinuation of the medication before 24 weeks by the clinical team or patient will be considered a failure to tolerate the medicine.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 26
Participants | 3

3. Secondary Outcome: Number of Participants With Sustained Virologic Response
Description: Undetectable HDV RNA at both 12 and 24 weeks post treatment follow-up visits
Time Frame: 12 and 24 weeks after completing therapy
Population: 25 participants had data at 24 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 25
Participants | 3

4. Secondary Outcome: Number of Participants With Reduction in Histologic Inflammatory Scores (Modified HAI)
Description: Reduction in histologic inflammatory scores (modified HAI) by at least two points with no progression in histologic fibrosis (Ishak) at week 24 post-treatment follow-up.
Time Frame: End of treatment and 24 weeks after completing therapy.
Population: 21 participants had liver biopsies at 24 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 21
Participants | 6

5. Secondary Outcome: Number of Participants With Normalization of Serum ALT
Description: Normalization of serum ALT (ALT <20 in females and ALT <31 in males) at the end of therapy, at week 12 of posttherapy follow-up and at week 24 of post-therapy follow-up, OR reduction in serum ALT by >50% of baseline at week 12 of post therapy follow up and week 24 of post therapy follow up.
Time Frame: End of therapy, and 12 and 24 weeks after completing therapy
Population: Two participants did not have ALT measures at 12 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 24
Participants | 2

6. Secondary Outcome: Number of Participants With Reduction of Hepatic Venous Pressure Gradient (HVPG)
Description: Reduction in hepatic venous pressure gradient (HVPG) measurements by >25% of baseline OR normalization of HVPG (<5 mm Hg) at 24 weeks after completing therapy
Time Frame: Baseline and 24 weeks after completing therapy
Population: Five participant did not have HVPG measured at 24 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 21
Participants | 10

7. Secondary Outcome: Number of Participants With Reduction in Fibroscan Transient Elastography Values
Description: Reduction in Fibroscan transient elastography values by >25% of baseline at end of therapy.
Time Frame: Baseline and 24 weeks
Population: Only 13 participants had Fibroscans at baseline and 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 13
Participants | 4

8. Secondary Outcome: Number of Participants With Loss of HBsAg at Week 24
Description: Loss of HBsAg from the serum at week 24
Time Frame: Week 24
Population: 22 participants had HBsAg values at week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 22
Participants | 0

9. Secondary Outcome: Number of Participants With Loss of HBsAg at Week 12 Weeks After Completing Therapy
Description: Loss of HBsAg from the serum at 12 weeks after completing therapy
Time Frame: 12 weeks after completing therapy
Population: 24 participants had HBsAg measurements at 12 weeks after the end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 24
Participants | 0

10. Secondary Outcome: Number of Participants With Loss of HBsAg at 24 Weeks After Completing Therapy
Description: Loss of HBsAg from the serum at 24 weeks after completing therapy
Time Frame: 24 weeks after completing therapy
Population: 24 participants had HBsAg measurements at 24 weeks after the end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 24
Participants | 0

11. Secondary Outcome: Change in Quantitative Log HBsAg Levels From Baseline to Week 24
Description: Change in quantitative log HBsAg levels at from baseline to week 24
Time Frame: Baseline and week 24
Population: 22 participants had HBsAg values at week 24
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Treatment
Number analyzed (Participants) | 22
log IU/mL | 0.15 (0.22)

12. Secondary Outcome: Change in Quantitative Log HBsAg Levels From Baseline 24 Weeks After Completing Therapy
Description: Change in quantitative log HBsAg levels at from baseline to 24 weeks after completing therapy
Time Frame: Baseline and 24 weeks after completing therapy
Population: 24 participants had HBsAg measurements at 24 weeks after the end of treatment
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Treatment
Number analyzed (Participants) | 24
log IU/mL | 0.16 (0.19)

ADVERSE EVENTS:
Time Frame: 48 Weeks
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 24/26
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=26)
Nausea (Gastrointestinal disorders) | 18
Diarrhea (Gastrointestinal disorders) | 21
Decreased Appetite (Metabolism and nutrition disorders) | 13
GERD (Gastrointestinal disorders) | 15
Fatigue (Musculoskeletal and connective tissue disorders) | 8
Headache (Nervous system disorders) | 1
Weight Loss (Investigations) | 6
Acneiform Rash (Skin and subcutaneous tissue disorders) | 4
Hyperbilirubinemia (Hepatobiliary disorders) | 6
Ascites (Hepatobiliary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Insomnia (Nervous system disorders) | 2
Hair Loss (Skin and subcutaneous tissue disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT03600714/Prot_SAP_000.pdf